CLINICAL TRIAL: NCT02577484
Title: Assessment of Catheter-based Interrogation and Standard Techniques for Fractional Flow Reserve Measurement: the ACIST-FFR Study
Brief Title: Assessment of Catheter-based Interrogation and Standard Techniques for Fractional Flow Reserve Measurement
Acronym: ACIST-FFR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Acist Medical Systems (Industry)
Responsible Party: Sponsor
Other Study IDs: US100
Record Dates: First submitted 2015-10-13; First posted 2015-10-16 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Disease
Keywords: Fractional Flow Reserve; Rapid Exchange; Catheter
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants: Subjects who satisfy both general and angiographic inclusion/exclusion criteria, and who have the pressure measurement taken with the Navvus catheter.
  Interventions: Device: RXi System; Device: Pressure Wire

INTERVENTIONS:
Device: RXi System — Provide hemodynamic information for the diagnosis and treatment of coronary and peripheral artery disease. The system is intended for use in catheterization and related cardiovascular specialty laboratories to compute and display fractional flow reserve or FFR.
  Measurement of FFR requires simultaneously monitoring the blood pressures proximal and distal to a lesion. The RXi system includes a single use catheter (Navvus) with a pressure sensor for acquisition of the distal pressure. The proximal pressure is acquired by the guide catheter via an interface to the hospital hemodynamic monitor.
  The Navvus catheter interfaces to the RXi system console which includes embedded software, a user interface touch screen and associated electronics.
  Other Names: ACIST Medical Systems RXi System; Navvus Catheter
Device: Pressure Wire — Provide hemodynamic information for the diagnosis and treatment of coronary and peripheral artery disease. The system is intended for use in catheterization and related cardiovascular specialty laboratories to compute and display fractional flow reserve or FFR.
  Other Names: St. Jude PressueWire Aeris Guidewire; St. Jude PressureWire Certus Guidewire; Volcano PrimeWire Prestige

SUMMARY:
This study will assess the differences between Fractional Flow Reserve (FFR) measurements made by the Navvus catheter and a commercially available pressure guidewire in up to 240 subjects where FFR is clinically indicated. All subjects will receive diagnostic treatment according to clinical indications and center standard practice.

DETAILED DESCRIPTION:
The ACIST-FFR study is a prospective, open label, observational, multi-center study designed to assess the differences, if any, between FFR measured by the Navvus catheter and a commercially available 0.014-inch pressure guidewire (St. Jude Medical, Volcano, hereafter referred to as the PW) in subjects with coronary artery disease (CAD) undergoing coronary angiography. This will be accomplished by comparing the FFR measurement obtained with the ACIST Medical Systems RXi System and Navvus catheter with the FFR measurement obtained by using a PW within the same subject across the same target lesion at the same time.

ELIGIBILITY:
General Inclusion Criteria:

* Subject is 18 years of age or older
* Subject has a clinical indication for coronary angiography
* Subject or subject's legal representative has the ability to understand and provide signed consent for participating in the study

Angiographic Inclusion Criteria:

* Vessel has a TIMI flow = 3
* Subject has de novo lesion which physician has determined has a clinical indication for FFR measurement
* RVD of the target lesion is assessed by the operator to be ≥2.25 mm.

General Exclusion Criteria:

* Subjects with acute ST-elevation or non-ST-elevation myocardial infarction as the indication for coronary angiography
* NYHA Class 4 severe heart failure

Angiographic Exclusion Criteria:

* Target vessel has angiographically visible or suspected thrombus.
* Target lesion is within a bypass graft.
* Angiographic evidence of a dissection prior to initiation of PW measurements.
* Target vessel contains excessive tortuosity or calcification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age or older, with single or multi-vessel CAD for whom FFR measurement is indicated to guide percutaneous coronary intervention strategy.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
FFR Measurements | Duration of FFR Procedure
  Bias between Navvus and PW FFR measurements, as assessed by Bland-Altman analysis

SECONDARY OUTCOMES:
Slope of Passing-Bablok | Duration of FFR Procedure
  Slope of Passing-Bablok fit between paired FFR measurements by Navvus and PW
Intercept of Passing-Bablok | Duration of FFR Procedure
  Intercept of Passing-Bablok fit between paired FFR measurements by Navvus and PW
Comparability of FFR Measurements | Duration of FFR Procedure
  Comparability of PW FFR and Navvus FFR measurements at PW FFR=0.80, by Passing-Bablok analysis.
Diagnostic FFR concurrence of stenosis significance | Duration of FFR Procedure
  Concurrence of Navvus FFR diagnostic accuracy of stenosis significance, using PW FFR ≤0.80 as the standard.
Device success rate | Duration of FFR Procedure
  Device success rate, defined as a valid FFR reading, for each system individually, and comparison between the two systems.
Mean drift | Duration of FFR Procedure
  Mean drift, defined as the absolute difference between Pd/Pa at the equalization position after pullback and 1.00, for each system individually, and comparison between the two systems.
Rate of clinically significant drift | Duration of FFR Procedure
  Rate of clinically significant drift, defined as drift >0.03, for each system individually, and comparison between the two systems.
Rate of device-related adverse effects | Duration of FFR Procedure
  Rate of device-related adverse effects, for each system individually, and comparison between the two systems.
PW FFR measurements with Navvus across and not across lesion | Duration of FFR Procedure
  Comparisons between PW FFR measurements with Navvus across lesion and with Navvus not across lesion, including bias as assessed by Bland-Altman analysis.
Comparison of FFR Measurements including bias | Duration of FFR Procedure
  Comparisons between PW (with Navvus present in lesion) and Navvus FFR measurements, including bias assessed by Bland-Altman analysis.
Correlation between Navvus diagnostic accuracy, bias, and angiographic characteristics | Duration of FFR Procedure
  Relationship between Navvus diagnostic accuracy, bias, and angiographic characteristics such as lesion length and reference vessel diameter.
PW Pd/Pa diagnostic concurrence of stenosis signficance | Duration of FFR Procedure
  PW Pd/Pa diagnostic accuracy (concurrence) of stenosis significance, using PW FFR ≤0.80 as the standard.
PW Pd/Pa measurements with Navvus across and not across lesion | Duration of FFR Procedure
  Comparisons between PW Pd/Pa measurements with Navvus across lesion and with Navvus not across lesion, including bias as assessed by Bland-Altman analysis.
Comparison of Pd/Pa Measurements including bias | Duration of FFR Procedure
  Comparisons between PW (with Navvus present in lesion) and Navvus Pd/Pa measurements, including bias assessed by Bland-Altman analysis.

CONTACTS AND LOCATIONS:
Overall Officials: William Fearon, MD, Principal Investigator — Stanford Cardiovascular Medical Clinic; Matthew Price, MD, Principal Investigator — Scripps Green Hospital
Locations (12):
- United States (12):
  - Scripps Green Hospital, La Jolla, California
  - Long Beach VA Medical Center, Long Beach, California
  - Stanford School of Medicine, Stanford, California
  - Medstart Washington Hospital Center, Washington D.C., District of Columbia
  - University of Chicago Medicine, Chicago, Illinois
  - Iowa Heart Center, West Des Moines, Iowa
  - Metropolitan Cardiology Heart and Vascular Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Columbia University Medical Center / New York Presbyterian Hospital, New York, New York
  - Lindner Research Center at The Christ Hospital, Cincinnati, Ohio
  - Cleveland Cllinic Foundation, Cleveland, Ohio

REFERENCES:
- [Background] Fearon WF, Bornschein B, Tonino PA, Gothe RM, Bruyne BD, Pijls NH, Siebert U; Fractional Flow Reserve Versus Angiography for Multivessel Evaluation (FAME) Study Investigators. Economic evaluation of fractional flow reserve-guided percutaneous coronary intervention in patients with multivessel disease. Circulation. 2010 Dec 14;122(24):2545-50. doi: 10.1161/CIRCULATIONAHA.109.925396. Epub 2010 Nov 29. PMID 21126973
- [Background] Fearon WF, Tonino PA, De Bruyne B, Siebert U, Pijls NH; FAME Study Investigators. Rationale and design of the Fractional Flow Reserve versus Angiography for Multivessel Evaluation (FAME) study. Am Heart J. 2007 Oct;154(4):632-6. doi: 10.1016/j.ahj.2007.06.012. PMID 17892983
- [Background] King SB 3rd, Smith SC Jr, Hirshfeld JW Jr, Jacobs AK, Morrison DA, Williams DO, Feldman TE, Kern MJ, O'Neill WW, Schaff HV, Whitlow PL; ACC/AHA/SCAI; Adams CD, Anderson JL, Buller CE, Creager MA, Ettinger SM, Halperin JL, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura R, Page RL, Riegel B, Tarkington LG, Yancy CW. 2007 focused update of the ACC/AHA/SCAI 2005 guideline update for percutaneous coronary intervention: a report of the American College of Cardiology/American Heart Association Task Force on Practice guidelines. J Am Coll Cardiol. 2008 Jan 15;51(2):172-209. doi: 10.1016/j.jacc.2007.10.002. No abstract available. PMID 18191745
- [Background] Pijls NH, Fearon WF, Tonino PA, Siebert U, Ikeno F, Bornschein B, van't Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, De Bruyne B; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention in patients with multivessel coronary artery disease: 2-year follow-up of the FAME (Fractional Flow Reserve Versus Angiography for Multivessel Evaluation) study. J Am Coll Cardiol. 2010 Jul 13;56(3):177-84. doi: 10.1016/j.jacc.2010.04.012. Epub 2010 May 28. PMID 20537493
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Derived] Fearon WF, Chambers JW, Seto AH, Sarembock IJ, Raveendran G, Sakarovitch C, Yang L, Desai M, Jeremias A, Price MJ; ACIST-FFR Study Investigators. ACIST-FFR Study (Assessment of Catheter-Based Interrogation and Standard Techniques for Fractional Flow Reserve Measurement). Circ Cardiovasc Interv. 2017 Dec;10(12):e005905. doi: 10.1161/CIRCINTERVENTIONS.117.005905. PMID 29246917